CLINICAL TRIAL: NCT00684840
Title: Biobehavioral Study of Opioid Drug Seeking Behavior: Study 4
Brief Title: Effects of Stress and Other Factors on Opiate Drug Choice.
Acronym: DSS
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Principal Investigator, Wayne State University
Other Study IDs: NIDA-15462-4; R01DA015462-04 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Behavioral Economics; Drug self administration; Opioid
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose is to study the extent to which stress and other factors, including money, the amount of drug available and the amount of work effort, affect drug choice.

This study will assess whether exposure to yohimbine, a drug stressor, increases opioid craving- and -seeking behavior. We will determine whether these behavioral outcomes are associated with biobehavioral stress markers: increased saliva cortisol levels, cardiovascular response (heart rate and blood pressure), and negative mood state.

DETAILED DESCRIPTION:
Physical, environmental, and pharmacological stressors have been repeatedly shown to increase self-administration of various abused substances in both preclinical and human studies. The primary aim of the proposed work is to assess the effects of yohimbine, a pharmacological agent, used to create an objectively-measured stress response, upon opioid-seeking behavior and craving.

Participants will first be an outpatient and must come to the Jefferson Avenue Research Program daily to receive buprenorphine doses. This phase will last at least 10 days or longer. Three times per week during the first two weeks (i.e., on 6 different days), participants will be asked to provide urine samples and to complete questionnaires that ask about opiate withdrawal symptoms.

Next, participants will live on an inpatient research unit for at least 11 consecutive nights and possibly up to 15 consecutive nights. During this stay they will participate in a total of eight experimental sessions. Participants will take part in multiple trials in which they have the opportunity to choose drug, hydromorphone (HYD), or money. HYD is a drug that is currently used as a cough suppressant and to relieve pain. During the first two test sessions, participants will receive a sample of the drug doses that can be chosen. Before each of the final 6 test sessions begin, participants will be given a capsule containing either different doses of the drug yohimbine or a placebo (blank). Yohimbine is a drug that has been shown to produce a "stress"-like response in humans. Then participants will have 12 opportunities to choose either drug or money by using a computer to earn choices. Respiration rate, oxygen saturation, heart rate, and blood pressure will be monitored throughout choice trials. Self-report questionnaires will be completed at different times during the study.

After participants have completed the experimental procedures, they will again come to the Jefferson Ave. Research Program daily to receive buprenorphine doses. The dose of buprenorphine will be gradually decreased so that they will eventually be free from medication. This will take three weeks. We will administer questionnaires and collect urine samples three times each week to assess using illicit drugs.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependent, as determined by structured clinical interview for DSM-IV (SCID) and Addiction Severity Index (ASI)
* Positive urine test for opiates
* Willing to use an adequate form of contraception for the duration of the study.
* Reads and writes English

Exclusion Criteria:

* Psychiatric illness, as determined by the DSM-IV criteria
* History of or current neurological disease, including structural abnormalities, seizures, infection, peripheral neuropathy, and head traumas
* History of cardiovascular disease, myocardial infarction, chest pain, or edema
* Systolic blood pressure greater than 160mm HG or less than 95 mm HG: PR diastolic blood pressure greater than 95 mm HG.
* Pulmonary disease, including obstructive pulmonary disease, Cor pulmonale, tuberculosis, and asthma
* Systemic disease (e.g. endocrinopathies, liver or kidney failure, myxedema, hypothyroidism, Addison's disease, autoimmune disease)
* Current alcohol or sedative drug dependence
* Pregnant or breast feeding
* Currently receiving treatment for opioid dependence
* Known phobia of injections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Heroin dependent research volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Woodcock EA, Lundahl LH, Burmeister M, Greenwald MK. Functional mu opioid receptor polymorphism (OPRM1 A(118) G) associated with heroin use outcomes in Caucasian males: A pilot study. Am J Addict. 2015 Jun;24(4):329-35. doi: 10.1111/ajad.12187. Epub 2015 Apr 24. PMID 25911999
- [Derived] Stoltman JJ, Woodcock EA, Lister JJ, Greenwald MK, Lundahl LH. Exploration of the telescoping effect among not-in-treatment, intensive heroin-using research volunteers. Drug Alcohol Depend. 2015 Mar 1;148:217-20. doi: 10.1016/j.drugalcdep.2015.01.010. Epub 2015 Jan 19. PMID 25630964
- [Derived] Greenwald MK, Lundahl LH, Steinmiller CL. Yohimbine increases opioid-seeking behavior in heroin-dependent, buprenorphine-maintained individuals. Psychopharmacology (Berl). 2013 Feb;225(4):811-24. doi: 10.1007/s00213-012-2868-9. Epub 2012 Nov 17. PMID 23161001